CLINICAL TRIAL: NCT03865082
Title: Study of Tilsotolimod in Combination With Nivolumab and Ipilimumab for the Treatment of Solid Tumors
Brief Title: Study of Tilsotolimod in Combination With Nivolumab and Ipilimumab for the Treatment of Solid Tumors (ILLUMINATE-206)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2125-MST-206
Record Dates: First submitted 2019-02-08; First posted 2019-03-06 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — tilsotolimod; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IO Naive Subjects MSS CRC (Experimental): 8mg Tilsotolimod by intratumoral injection plus 3mg/kg Nivolumab (every three weeks for four doses followed by 480mg dose every four weeks) and 1mg/kg Ipilimumab every three weeks for four doses intravenous
  Interventions: Drug: Tilsotolimod; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Tilsotolimod — 9 doses of Tilsotolimod Intratumoral injection administered as a dose of 8mg at Week 0 Day 1 (7 days prior to the start of Cycle 1), Day 1 and Day 8 of Cycle 1, and on Day 1 of Cycles 2 through 7.
  Other Names: IMO-2125
Drug: Nivolumab — Specified dose on specified days.
  Other Names: OPDIVO
Drug: Ipilimumab — Specified dose on specified days.
  Other Names: Yervoy

SUMMARY:
A Phase 2 study intended to see efficacy of tilsotolimod in combination with immunotherapy drugs ipilimumab and nivolumab in different solid tumors.

DETAILED DESCRIPTION:
This is a Phase 2, open-label,multi-center, multicohort study of intratumoral tilsotolimod in combination with nivolumab and ipilimumab for the treatment of specific solid tumors

ELIGIBILITY:
Main Inclusion Criteria:

1. Subject must be willing and able to sign the informed consent and comply with study protocol.
2. Must be ≥ 18 years of age (males and females).
3. ≥ 1 lesion accessible for i.t. injection and biopsy(ies).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 minimum life expectancy ≥ 4 months.
5. Adequate baseline organ function as defined by:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500/mm3)
   2. Platelet count ≥ 100 x 109/L (100,000/mm3)
   3. Hemoglobin ≥ 9.0 g/dL (5.59 mmol/L)
   4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance of ≥ 40 mL/minute (measured or calculated using the Cockroft-Gault formula)
   5. Aspartate aminotransferase (AST) ≤ 3 x ULN, alanine aminotransferase (ALT) ≤ 3 x ULN; AST/ALT < 5 ULN if liver involvement
   6. ≤ 1.5 x ULN, except in subjects with Gilbert's syndrome who must have a total bilirubin ≤ 3 mg/dL
6. Women of child bearing potential (WOCBP) and men with WOCBP partners must agree to use effective contraception methods as defined in the clinical study protocol.
7. For any subjects who received prior approved/investigational i.t. anti-cancer treatments, the study's Medical Monitor must be consulted before enrollment.

Inclusion Criteria ( MSS CRC IO Naïve)

1. Histologically confirmed advanced, metastatic, or progressive MSS CRC based on either an analysis of tissue from a prior biopsy or based on tissue from a new biopsy. Subject's microsatellite/MMR status should be known.
2. Received two prior lines of therapy for advanced or metastatic CRC including fluoropyrimidine-, oxaliplatin-, and irinotecan-based regimens. Subjects who relapse within 6 months of adjuvant chemotherapy composed of oxaliplatin and a fluoropyrimidine will have their adjuvant therapy count as one prior regimen.
3. Documentation of radiologic progression by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 during or after previous chemotherapy. Subjects documented clinical progression may be eligible and must be discussed with the medical monitor to determine eligibility.

Main Exclusion Criteria:

1. Subject must have completed or completely discontinued any previous cancer-related treatments before enrollment with necessary windows and wash out periods as defined in the clinical study protocol.
2. History of interstitial lung disease, pneumonitis, known or suspected autoimmune diseases (unless for specific diseases as defined in protocol) or human immunodeficiency virus (HIV) infection.
3. Prior therapy with TLR9 agonist, excluding topical agents.
4. Known hypersensitivity to any study drug component.
5. Treatment with botanical preparations (e.g. herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to treatment.
6. Known or suspected autoimmune diseases. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to be enrolled.

   Subject with a requirement of systemic steroids > 10 mg/day of prednisone (or equivalent) for the 2 weeks preceding start of study treatment.
7. Subject with another primary malignancy that has not been in remission for at least 3 years except for non-melanoma skin cancer, curatively treated localized prostate cancer with non-detectable prostate specific antigen, cervical carcinoma in situ on biopsy, or thyroid cancer (except anaplastic).
8. Active systemic infections requiring antibiotics.
9. Active Hepatitis A, B or C infections.
10. Known diagnosis of human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS). NOTE: Testing for HIV must be performed at sites where mandated locally.
11. Women who are breast feeding or pregnant.
12. Prior anaphylactic or other severe infusion reaction associated with human antibody administration that cannot be managed by standard supportive measurements.
13. Presence of known central nervous system (CNS), meningeal, or epidural metastatic disease.However, subjects with known brain metastases are allowed if brain metastases are stable for≥ 4 weeks before the first dose of study treatment. Stable is defined as neurological symptoms not present or resolved at baseline, no radiological evidence of progression, and steroid requirement of prednisone ≤ 10 mg/day or equivalent.
14. Subject with unstable and impaired cardiac function or clinically significant cardiac disease per Investigator's clinical judgment.
15. Has received live attenuated vaccine 30 days before first study dose. Any live attenuated vaccine [e.g., varicella, zoster, yellow fever, rotavirus, oral polio and measles, mumps, rubella (MMR)] during treatment and until 100 days post last dose will be prohibited.

Exclusion Criteria (MSS CRC IO Naïve):

1. Prior therapy with an anti-programmed cell death-1 (PD-1), anti-programmed cell death ligand-1 (PD-L1), or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor in an approved or experimental setting.
2. Subjects with BRAF V600E mutations.
3. Subjects with a history of immune-mediated colitis.
4. Subjects who received three or more lines of therapy for advanced or metastatic CRC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-29 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the efficacy of intratumoral tilsotolimod in combination with ipilimumab and nivolumab for each cohort | ORR defined as a CR or partial response (PR) according to RECIST v1.1, confirmed by imaging ≥ 4 weeks after the initial documentation of response (to occur up to 24 months).
  Efficacy measure by objective response rate
Duration of response | DOR will be evaluated every 8 weeks starting Cycle3 Day1 (each cycle is 28 days) for year 1 then every 12 weeks after the first year through study completion until all study participants have either progressive disease or start new anticancer treatment.
  Durability or response per RECIST v1.1

SECONDARY OUTCOMES:
Safety and tolerability of the combination of tilsotolimod with nivolumab and ipilimumab | At every study visit (up to 48 months)
  Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms(ECGs), safety and laboratory parameters as assessed by CTCAE v4.03 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Idera Medical Director, Study Director — Idera Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Banner University Medical Center Tucson Campus, Tucson, Arizona
  - University of Southern California/ Hoag Hospital Presbyterian, Newport Beach, California
  - MD Anderson Cancer Center, Houston, Texas